CLINICAL TRIAL: NCT00505076
Title: MK-0777 for the Treatment of Cognitive Impairments in Patients With Schizophrenia
Brief Title: Treatment Study for Cognitive Deficits in Schizophrenia
Acronym: TURNS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of Maryland (Other); Washington University School of Medicine (Other); Massachusetts General Hospital (Other); Nathan Kline Institute for Psychiatric Research (Other); Columbia University (Other); Duke University (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Stephen R. Marder, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TURNS02; HHSN278200441003C (Other Grant/Funding Number: NIMH grant)
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Results first posted 2014-10-31 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Schizophrenia
Keywords: Cognition; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — 7-(1,1-dimethylethyl)-6-(2-ethyl-2H-1,2,4-triazol-3-ylmethoxy)-3-(2-fluorophenyl)-1,2,4-triazolo(4,3-b)pyridazine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MK-0777 8 mg (Experimental): MK-0777 8 mg tablet by mouth twice daily for 4 weeks
  Interventions: Drug: MK-0777
- MK-0777 3 mg (Experimental): MK-0777 3 mg tablet by mouth twice daily for 4 weeks
  Interventions: Drug: MK-0777
- Placebo (Placebo Comparator): Placebo tablet by mouth twice daily for 4 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: MK-0777 — MK-0777 GEM, 8 mg BID
  Arms: MK-0777 8 mg
Drug: MK-0777 — MK-0777 GEM, 3 mg BID
  Arms: MK-0777 3 mg
Drug: placebo — 2 tablets placebo BID
  Arms: Placebo

SUMMARY:
Patients with schizophrenia are characterized by a broad range of neurocognitive abnormalities. These include impairments in attention, including abnormalities in sensory gating; executive function; visual and verbal learning and memory; working memory; processing speed; and social cognition (Nuechterlein et al, 2004). These impairments are major determinants of poor functional outcome in patients with schizophrenia (Green, 1996; Green et al, 2004). Conventional antipsychotics have limited effects on these impairments. Second generation antipsychotics may have modest benefits for cognitive function, but whether this represents a direct cognitive enhancing effect has not been established. Regardless, patients continue to exhibit pronounced cognitive impairments despite adequate second generation antipsychotic treatment. Adjunctive pharmacotherapy may offer a viable approach for the treatment of cognitive impairments. Adjunctive agents can be used to modulate specific neurotransmitter systems that are hypothesized to be involved in the pharmacology of cognitive functions.

The standard of care for schizophrenia is antipsychotic medications to treat psychotic symptoms. However, cognitive impairments remain and these impairments have been found to be significantly associated with the poor psychosocial function observed in patients with schizophrenia. There is a considerable preclinical rationale for the use of drugs that act at the Gamma-amino-buyric acid (GABA) α2 subunit as adjunctive treatments to target cognitive impairments. MK-0777 GEM (Merck-0777 Gel Extrusion Module) formulation provides an opportunity to directly test this mechanism.

The purpose of the proposed study is to examine the efficacy and safety of two doses of MK (Merck) -0777 GEM, 3 mg BID (twice daily) and 8 mg BID (twice daily), in the treatment of cognitive impairments in patients with schizophrenia. Secondary goals are to determine whether MK-0777 has beneficial effects on measures of functional capacity and patient self-report of cognitive function.

DETAILED DESCRIPTION:
The proposed study is a multicenter, randomized, double blind comparison of MK-0777 GEM 3 mg BID, MK-0777 GEM 8 mg BID, and placebo. The total sample will consist of 90 clinically stable patients with DSM IV TR schizophrenia, with 30 subjects randomized to each group. A best estimate diagnostic approach will be utilized, in which information from the Structured Clinical Interview for DSM-IV (Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition) (First et al, 1997) is supplemented by information from family informants, previous psychiatrists, and medical records to generate a diagnosis. The projected number of subjects to be recruited from each site is 12-13. There will be a 2 week, placebo lead-in evaluation phase, in which subjects will undergo baseline diagnostic; medical, including a physical examination, EKG (electrocardiogram), CBC (Complete Blood Count), complete metabolic panel, urine toxicology, and UA (urinalysis); psychiatric; and neurocognitive, symptom level and functional capacity and patient self-report of cognitive function assessments. In addition, all subjects will receive a slit-lamp eye examination. At the end of the evaluation phase, subjects will be randomized to one of two MK-0777 doses or placebo. The double-blind treatment phase will be 4 weeks. Subjects will receive bi-weekly symptom assessments and weekly side effect and vital sign assessments. At week 4, subjects will undergo repeat administration of the neuropsychological test battery and the functional capacity and patient self-report of cognitive function measures. These assessments will be done over a two-day period. Subjects will have blood samples collected for antipsychotic and MK-0777 levels at week 4. An EKG (electrocardiogram) will be obtained at the end of the double-blind study. Slit-lamp eye examinations will be conducted at study completion, 6 months and 12 months after study completion. After the completion of the 4-week double-blind phase, there will be a 4-day follow-up phase during which subjects will be tapered off study medication.

Study Locations: The study will be conducted in the Treatment Units for Research on Neurocognition and Schizophrenia (TURNS) study network, which is comprised of seven sites: Columbia University School of Medicine (P.I.: Jeffrey Lieberman, M.D.); Duke University School of Medicine (P.I.: Joseph McEvoy, M.D.); Harvard University School of Medicine (P.I.: Donald Goff, M.D.); Maryland Psychiatric Research Center (MPRC) (P.I.: Robert W. Buchanan, M.D.); Nathan Kline Institute (P.I.: Daniel Javitt, M.D.) University of California Los Angeles School of Medicine (P.I.: Steve Marder, M.D.); and Washington University School of Medicine (P.I.: John Csernansky, M.D.). The TURNS is a NIMH-funded contract for the evaluation of new compounds for the treatment of cognitive impairments in schizophrenia (HHSN 27820044 1003C; P.I.: Steve Marder, M.D.). Data management will be performed by the Clinical Trials Data Management Unit of the Nathan Kline Institute under the direction of Jim Robinson, M.S., and statistical analysis will be performed by Dr. Robert McMahon of the Maryland Psychiatric Research Center. Laboratory assays will be performed by Quest Diagnostics.

Procedures:

Clinical Assessments: The symptom assessments will include the Brief Psychiatric Rating Scale; Scale for the Assessment of Negative Symptoms (SANS); Calgary Depression Scale (CDS); and Clinical Global Impression Scale (CGI).

i) BPRS(Brief Psychiatric Rating Scale): the four positive symptom items (conceptual disorganization, suspiciousness, hallucinatory behavior, and unusual thought content) will be used to measure positive psychotic symptoms.

ii) SANS (Scale for Assessment of Negative Symptoms): the SANS total score, minus the global items, inappropriate affect, poverty of content of speech, and attention items, will be used to measure negative symptoms. The inappropriate affect, poverty of content of speech, and attention items are excluded as lacking construct validity and because factor analytic study results suggest that these items are not closely related to negative symptoms.

iii) CDS (Calgary Depression Scale): the CDS total score will be used to measure depressive symptoms.

iv) CGI (Clinical Global Impressions): the CGI severity of illness item will be used to assess global changes

Safety Assessments: The safety assessments will include the Simpson Angus Extrapyramidal Symptom Rating Scale (SAS); Abnormal Involuntary Movement Scale (AIMS); and Side Effect Checklist (SEC).

i) SAS: a modified 11 item version of the SAS will be used to assess EPS. ii) AIMS: is a 12 item scale, with 7 items designed to assess abnormal facial, oral, extremity, and trunk movements; 3 global judgment items; and 2 current dental status items.

iii) SEC: is designed to assess vital signs, commonly occurring antipsychotic side effects, and side effects indicative of uveitis or cataracts.

Subjects will be asked about adverse events at each visit, and instructed to call the study site should they experience adverse events at any point in the study. Any serious adverse event, including death due to any cause, which occurs to any subject entered into this study or within 14 days following cessation of treatment, whether or not related to the investigational product, will be reported to Merck & Co., Inc. within 24 hours.

Functional Assessments: The functional assessments will include the UCSD Performance-Based Skills Assessment (UPSA) and the Schizophrenia Cognition Rating Scale (SCoRS).

i) UPSA: is designed to assess skills in five areas: household chores, communication, finance, transportation, and planning recreational activities. Subjects are asked to perform tasks in each of these areas and scored according to their ability to complete the task. The UPSA takes 25 - 30 minutes to administer.

ii) SCoRS: is a rating scale designed to elicit information from the subject and informant on the level of cognitive function of the subject. The subject and informant versions both have 20 items. Subject and informant interviews take from 10 - 15 minutes to complete.

Neurocognitive Assessments: The NIMH MATRICS (Measurement and Treatment Research to Improve Cognition in Schizophrenia Research) Neuropsychological Battery, the Wechsler Test of Adult Reading (WTAR), the N-Back test; and the Continuous Performance Test (CPT-AX) will be used to assess cognitive function. The NIMH MATRICS Neuropsychological Battery is comprised of measures of: a) working memory; b) attention/vigilance; c) verbal memory; d) visual memory; e) processing speed; f) problem solving; and g) social cognition. The N-Back and CPT-AX are both computerized measures of prefrontal cortex dependent cognitive behavior.

Screening: The diagnosis of schizophrenia will be confirmed by a research psychiatrist using a modified version of the Structured Clinical Interview for DSM IV (SCID). The BPRS, SANS, CDRS and SAS will be administered to verify that inclusionary criteria are met. Subjects will have a slit-lamp eye examination.

2 Week, Lead-in Evaluation Phase: In the 2 week lead-in evaluation phase, subjects will receive placebo. They will undergo baseline symptom, medical, safety, and neurocognitive assessments. The subjects will undergo a physical examination; including neurological exam, an EKG; and laboratory tests of major organ functions (i.e., CBC (complete blood count), liver function tests, electrolytes, glucose, BUN/Creatinine, Urinalysis (UA), urine toxicology, and thyroid functions). Baseline antipsychotic levels will be collected. All women will have a pregnancy test, unless they are either surgically or hormonally post menopausal.

4-Week Double Blind Treatment Phase: The study is a 4-week, placebo controlled, double blind study. Subjects will be randomized to either: MK-0777 GEM 3mg BID; MK-0777 GEM 8mg BID; or placebo. The unblinded site pharmacist will be notified of the treatment assignment, and will dispense study medication. Subjects will receive biweekly symptom assessments and weekly side effect and vital sign assessments. At week 4, subjects will undergo repeat administration of the neuropsychological test battery and the functional capacity and patient self-report of cognitive function measures. These assessments will be done over a two-day period. At week 4, subjects will also undergo a repeat slit lamp eye examination. We will also attempt to contact and schedule subjects who dropped out of the study prior to week 4 for the week 4 slit lamp eye examination. Finally, subjects will have blood samples collected for antipsychotic and MK-0777 levels at week 4.

6-Month and 12-Month Follow-up Evaluations: All subjects, regardless if they completed the 4-week double-blind treatment phase, will be contacted and scheduled for follow-up slit lamp eye examinations.

Randomization: Subjects will be randomly assigned to placebo or one of two doses of experimental treatment within strata defined by site.

Recruitment: Recruitment for potential subjects will be performed by reviewing subject records to determine eligibility based on the inclusion and exclusion criteria. Once qualifying records have been identified, potential subjects will be informed individually and/or in a group setting about the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: DSM IV/DSM IV TR schizophrenia (including disorganized, paranoid, undifferentiated, and catatonic subtypes)
* Capable of providing informed consent
* Duration of illness equal to or greater than one year
* Treated with one or two of the following second generation antipsychotics: risperidone, paliperidone, olanzapine, quetiapine, ziprasidone, or aripiprazole for the previous two months, with no change in dose in the last month.
* Meet the following symptom criteria:

  * Brief Psychiatric Rating Scale (BPRS) Hallucinatory Behavior, Unusual Thought Content or Conceptual Disorganization item score ≤ 4
  * All Scale for the Assessment of Negative Symptoms global items ≤ 3
  * Simpson-Angus Scale total score ≤ 6
  * Calgary Depression Scale total score ≤ 10
* Meet the following cognitive performance criteria:

  * Performance less than the maximum cutoff (in parentheses) for ONE of the following MCCB tests: i.) Letter-number span (20); ii.) HVLT total (31); and iii.) CPT d-prime (3.47)
  * Able to complete the baseline MCCB validly
  * Raw score ≥6 on the WTAR

Exclusion Criteria:

* Current treatment (within 4 weeks) with conventional antipsychotics (e.g. fluphenazine, haloperidol) or clozapine
* Current treatment with psychotropic agents known to act at the GABAA receptor, including benzodiazepines; sedative-hypnotics other than trazadone and chloral hydrate; carbamazepine, gabapentin, lamotrigine, and valproic acid
* Current treatment with a drug that inhibits CYP3A4, including: cimetidine; cyclosporine; erythromycin or erythromycin-like drugs (e.g., azithromycin, clarithromycin); diltiazem; fluoxetine, fluovoxamine; itraconazole, ketoconazole or other systemic antifungal agents in the azole class; nefazodone; or induce CYP3A4, including: carbamazepine, modafinil; phenobarbital; phenytoin; rifampin; St. Johns wort; and troglitazone.
* Current treatment with psychotropic agents known to effect cognition: amphetamine; barbiturates; lithium; MAOIs; methylphenidate
* Current treatment with herbal preparations with possible psychotropic effects (e.g., St. Johns wort, kava-kava, Valerian, S-Adenosyl Methionine [SAMe])
* Current treatment with systemic steroids
* DSM-IV diagnosis of alcohol or substance abuse (other than nicotine) within the last month or a DSM-IV diagnosis of alcohol or substance dependence within the last 6 months
* Presence of PI or greater posterior subcapsular cataracts
* Uveitis with 1+ or greater flare or cells
* Nuclear or cortical cataracts
* History of significant head injury/trauma, as defined by one or more of the following: loss of consciousness (LOC) for more than 1 hour, seizures from the head injury, clear cognitive sequellae of the injury, or cognitive rehabilitation following the injury
* History of clinically significant neurological, metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, and/or urological disorders.
* Clinically significant abnormalities in physical examination, ECG, or laboratory assessments
* A positive test for Hepatitis C antibody with concurrent evidence of impaired hepatic function (increased AST or ALT greater than 2 times the upper limit of normal) or positive tests for Hepatitis A antibody IgM fraction or Hepatitis B surface antigen, irrespective of the AST or ALT values.
* Pregnant women or women of child-bearing potential, either not surgically-sterile or using appropriate methods of birth control
* Women who are breast-feeding
* History of severe symptoms of benzodiazepine withdrawal (e.g., history of seizures or delirium associated with withdrawal)
* Received ECT treatment within the last 3 months
* Participated in a clinical trial of any other psychotropic medication within 2 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2007-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Buchanan, M.D., Principal Investigator — Maryland Psychiatric Research Center
Locations (8):
- United States (8):
  - UCLA, Los Angeles, California
  - Maryland Psychiatric Research Center, Catonsville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Harvard Medical School, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Nathan Kline Institute, Orangeburg, New York
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Background] Akbarian S, Kim JJ, Potkin SG, Hagman JO, Tafazzoli A, Bunney WE Jr, Jones EG. Gene expression for glutamic acid decarboxylase is reduced without loss of neurons in prefrontal cortex of schizophrenics. Arch Gen Psychiatry. 1995 Apr;52(4):258-66. doi: 10.1001/archpsyc.1995.03950160008002. PMID 7702443
- [Background] Callicott JH, Mattay VS, Bertolino A, Finn K, Coppola R, Frank JA, Goldberg TE, Weinberger DR. Physiological characteristics of capacity constraints in working memory as revealed by functional MRI. Cereb Cortex. 1999 Jan-Feb;9(1):20-6. doi: 10.1093/cercor/9.1.20. PMID 10022492
- [Background] Callicott JH, Ramsey NF, Tallent K, Bertolino A, Knable MB, Coppola R, Goldberg T, van Gelderen P, Mattay VS, Frank JA, Moonen CT, Weinberger DR. Functional magnetic resonance imaging brain mapping in psychiatry: methodological issues illustrated in a study of working memory in schizophrenia. Neuropsychopharmacology. 1998 Mar;18(3):186-96. doi: 10.1016/S0893-133X(97)00096-1. PMID 9471116
- [Background] Carpenter WT Jr, Buchanan RW, Kirkpatrick B, Breier AF. Diazepam treatment of early signs of exacerbation in schizophrenia. Am J Psychiatry. 1999 Feb;156(2):299-303. doi: 10.1176/ajp.156.2.299. PMID 9989567
- [Background] Carter CS, Perlstein W, Ganguli R, Brar J, Mintun M, Cohen JD. Functional hypofrontality and working memory dysfunction in schizophrenia. Am J Psychiatry. 1998 Sep;155(9):1285-7. doi: 10.1176/ajp.155.9.1285. PMID 9734557
- [Background] Gold JM, Carpenter C, Randolph C, Goldberg TE, Weinberger DR. Auditory working memory and Wisconsin Card Sorting Test performance in schizophrenia. Arch Gen Psychiatry. 1997 Feb;54(2):159-65. doi: 10.1001/archpsyc.1997.01830140071013. PMID 9040284
- [Background] Green MF. What are the functional consequences of neurocognitive deficits in schizophrenia? Am J Psychiatry. 1996 Mar;153(3):321-30. doi: 10.1176/ajp.153.3.321. PMID 8610818
- [Background] Green MF, Kern RS, Heaton RK. Longitudinal studies of cognition and functional outcome in schizophrenia: implications for MATRICS. Schizophr Res. 2004 Dec 15;72(1):41-51. doi: 10.1016/j.schres.2004.09.009. PMID 15531406
- [Background] Guidotti A, Auta J, Davis JM, Di-Giorgi-Gerevini V, Dwivedi Y, Grayson DR, Impagnatiello F, Pandey G, Pesold C, Sharma R, Uzunov D, Costa E. Decrease in reelin and glutamic acid decarboxylase67 (GAD67) expression in schizophrenia and bipolar disorder: a postmortem brain study. Arch Gen Psychiatry. 2000 Nov;57(11):1061-9. doi: 10.1001/archpsyc.57.11.1061. PMID 11074872
- [Background] Hashimoto T, Volk DW, Eggan SM, Mirnics K, Pierri JN, Sun Z, Sampson AR, Lewis DA. Gene expression deficits in a subclass of GABA neurons in the prefrontal cortex of subjects with schizophrenia. J Neurosci. 2003 Jul 16;23(15):6315-26. doi: 10.1523/JNEUROSCI.23-15-06315.2003. PMID 12867516
- [Background] Lewis DA, Hashimoto T, Volk DW. Cortical inhibitory neurons and schizophrenia. Nat Rev Neurosci. 2005 Apr;6(4):312-24. doi: 10.1038/nrn1648. PMID 15803162
- [Background] McMahon RP, Arndt S, Conley RR. More powerful two-sample tests for differences in repeated measures of adverse effects in psychiatric trials when only some patients may be at risk. Stat Med. 2005 Jan 15;24(1):11-21. doi: 10.1002/sim.1837. PMID 15515151
- [Background] Mirnics K, Middleton FA, Marquez A, Lewis DA, Levitt P. Molecular characterization of schizophrenia viewed by microarray analysis of gene expression in prefrontal cortex. Neuron. 2000 Oct;28(1):53-67. doi: 10.1016/s0896-6273(00)00085-4. PMID 11086983
- [Background] Nuechterlein KH, Barch DM, Gold JM, Goldberg TE, Green MF, Heaton RK. Identification of separable cognitive factors in schizophrenia. Schizophr Res. 2004 Dec 15;72(1):29-39. doi: 10.1016/j.schres.2004.09.007. PMID 15531405
- [Background] Park S, Holzman PS. Schizophrenics show spatial working memory deficits. Arch Gen Psychiatry. 1992 Dec;49(12):975-82. doi: 10.1001/archpsyc.1992.01820120063009. PMID 1449384
- [Background] Pierri JN, Chaudry AS, Woo TU, Lewis DA. Alterations in chandelier neuron axon terminals in the prefrontal cortex of schizophrenic subjects. Am J Psychiatry. 1999 Nov;156(11):1709-19. doi: 10.1176/ajp.156.11.1709. PMID 10553733
- [Background] Rao SG, Williams GV, Goldman-Rakic PS. Isodirectional tuning of adjacent interneurons and pyramidal cells during working memory: evidence for microcolumnar organization in PFC. J Neurophysiol. 1999 Apr;81(4):1903-16. doi: 10.1152/jn.1999.81.4.1903. PMID 10200225
- [Background] Rao SG, Williams GV, Goldman-Rakic PS. Destruction and creation of spatial tuning by disinhibition: GABA(A) blockade of prefrontal cortical neurons engaged by working memory. J Neurosci. 2000 Jan 1;20(1):485-94. doi: 10.1523/JNEUROSCI.20-01-00485.2000. PMID 10627624
- [Derived] Georgiades A, Davis VG, Atkins AS, Khan A, Walker TW, Loebel A, Haig G, Hilt DC, Dunayevich E, Umbricht D, Sand M, Keefe RSE. Psychometric characteristics of the MATRICS Consensus Cognitive Battery in a large pooled cohort of stable schizophrenia patients. Schizophr Res. 2017 Dec;190:172-179. doi: 10.1016/j.schres.2017.03.040. Epub 2017 Apr 20. PMID 28433500
- [Derived] Buchanan RW, Keefe RS, Lieberman JA, Barch DM, Csernansky JG, Goff DC, Gold JM, Green MF, Jarskog LF, Javitt DC, Kimhy D, Kraus MS, McEvoy JP, Mesholam-Gately RI, Seidman LJ, Ball MP, McMahon RP, Kern RS, Robinson J, Marder SR. A randomized clinical trial of MK-0777 for the treatment of cognitive impairments in people with schizophrenia. Biol Psychiatry. 2011 Mar 1;69(5):442-9. doi: 10.1016/j.biopsych.2010.09.052. Epub 2010 Dec 8. PMID 21145041

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between June 2007 and July 2009.
Pre-assignment Details: 46 subjects were excluded during screening.
Groups:
- MK-0777 8 mg BID: Subjects treated with MK-0777 GEM, 8 mg BID(twice daily)
- MK-0777 3 mg BID: Subjects treated with MK-0777 GEM, 3 mg BID (twice daily)
- Placebo BID: Subjects treated with 2 tablets placebo BID (twice daily)
Period: Overall Study
Arm/Group | MK-0777 8 mg BID | MK-0777 3 mg BID | Placebo BID
Started | 22 | 19 | 22
Completed | 19 | 17 | 17
Not Completed | 3 | 2 | 5
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Protocol Violation | 2 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- MK-077 8 mg BID: Subjects treated with MK-0777 GEM, 8 mg BID(twice daily)
- Total: Total of all reporting groups
Arm/Group | MK-077 8 mg BID | MK-0777 3 mg BID | Placebo BID | Total
Number analyzed (Participants) | 22 | 19 | 22 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 19 | 22 | 63
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (8.7) | 43.3 (9.3) | 40.0 (10.9) | 42.7 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 6 | 23
  Male | 13 | 11 | 16 | 40
Region of Enrollment [Number; unit: participants]
  United States | 22 | 19 | 22 | 63

OUTCOME MEASURES:

1. Primary Outcome: Composite MATRICS Consensus Cognitive Battery Score
Description: The primary outcome measure is the composite score on the Matrics Consensus Cognitive Battery (MCCB). The MCCB composite score is a standardized mean of the seven domain scores. T-scores are standardized to normative data, and have an estimated mean of 50 and SD of 10 in the general healthy population. Data reduction for analysis of neurocognitive testing used the following steps: i) individual neurocognitive test scores at baseline and follow-up were converted to t-scores; ii) t-scores within the pre-specified cognitive domains measured by more than one test were averaged to obtain a domain-specific t-score; and iii) domain-specific t-scores were averaged to create the MCCB composite score.
Time Frame: 4 weeks
Population: Fifty-three participants completed the study: MK-0777 3mg BID: 18; MK-0777 8mg BID: 18; placebo: 17. Three participants dropped out prior to receiving study drug (one randomized to each group) and 1 participant dropped out prior to any post-randomization ratings (randomized to placebo). These participants were not included in analyses.
Measure: Mean (Standard Deviation); unit: composite score
Groups:
- MK-077 8 mg BID: Subjects treated with MK-0777, 8 mg BID
- MK-0777 3 mg BID: Subjects treated with MK-0777 , 3 mg BID
- Placebo BID: Subjects treated with placebo tablet BID
Arm/Group | MK-077 8 mg BID | MK-0777 3 mg BID | Placebo BID
Number analyzed (Participants) | 18 | 18 | 17
composite score | 27.9 (12.7) | 31.3 (13.9) | 32.5 (14.0)
Statistical Analysis 1: Comparison: MK-077 8 mg BID vs MK-0777 3 mg BID vs Placebo BID; An analysis of covariance (ANCOVA), adjusting for baseline scores, was used to compare treatment groups on cognitive and functional measures. The predefined primary cognition outcome measure was the MCCB (MATRICS (Measurement and Treatment Research to Improve Cognition in Schizophrenia Research) Consensus Cognitive Battery) composite T-score, tested at overall two-sided alpha=0.05; Test type: Superiority or Other; p = 0.21, ANCOVA

2. Secondary Outcome: UPSA(UCSD Performance-Based Skills Assessment) Summary Score
Description: The UCSD Performance-Based Skills Assessment assessed functional capacity. The UPSA Summary Score has a range from 0 to 120. A higher score indicates less impairment.
Time Frame: Baseline and end of treatment, a total of four weeks.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: UPSA Summary Score
Arm/Group | MK-077 8 mg BID | MK-0777 3 mg BID | Placebo BID
Number analyzed (Participants) | 18 | 18 | 17
UPSA Summary Score
  Baseline | 91.7 (13.4) | 85.0 (18.8) | 95.0 (16.3)
  End of Treatment | 90.4 (12.8) | 86.3 (18.7) | 96.5 (15.5)
Statistical Analysis 1: Comparison: MK-077 8 mg BID vs MK-0777 3 mg BID vs Placebo BID; The sample size was determined using the analysis of covariance power formula, n=2[za+zβ]2s2 (1-R2)/d2, with za=2.24, zβ=0.842 (corresponding to power=0.80), R=the correlation between baseline and end of study measures of the outcome, d the difference between groups, and s the standard deviation of the outcome. Actual recruitment was only about 20 participants per group, but the observed R≅0.9, suggesting power to detect an effect size of 0.49; Test type: Superiority or Other; p = 0.47, ANCOVA

3. Secondary Outcome: Schizophrenia Cognition Rating Scale (SCoRS) Score
Description: The Schizophrenia Cognition Rating Scale (SCoRS) assessed functional capacity. The SCoRS Interviewer Global Rating of function has a range 1 to 10. Higher ratings indicate greater impairment.
Time Frame: 4 Weeks (Baseline to End of Treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SCoRS Score
Arm/Group | MK-077 8 mg BID | MK-0777 3 mg BID | Placebo BID
Number analyzed (Participants) | 18 | 18 | 17
SCoRS Score
  Baseline | 4.1 (2.3) | 4.8 (2.3) | 3.8 (2.3)
  End of Treatment | 4.0 (2.4) | 4.6 (2.1) | 3.6 (1.8)
Statistical Analysis 1: Comparison: MK-077 8 mg BID vs MK-0777 3 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.84, ANCOVA

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | MK-077 8 mg BID | MK-0777 3 mg BID | Placebo BID
Serious Adverse Events (participants affected / at risk) | 1/21 | 1/18 | 0/21
Other Adverse Events (participants affected / at risk) | 7/21 | 2/18 | 5/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-077 8 mg BID (N=21) | MK-0777 3 mg BID (N=18) | Placebo BID (N=21)
Medical Hospitalization (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Fever with influenza
Psychosis Hospitalization (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Hospitalization for psychosis
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-077 8 mg BID (N=21) | MK-0777 3 mg BID (N=18) | Placebo BID (N=21)
Sedation (General disorders) | 2 (2) | 1 (1) | 1 (1)
Dizziness (General disorders) | 2 (2) | 0 (0) | 1 (1)
Fever (General disorders) | 2 (2) | 0 (0) | 0 (0)
Headache (General disorders) | 1 (1) | 0 (0) | 2 (2)
Limb pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No